CLINICAL TRIAL: NCT01443078
Title: Phase II Trial of Neoadjuvant Platinum-based Chemotherapy for Patients With Resectable , Non-small Cell Lung Cancer With Switch to Chemotherapy Alternative in Nonresponders (NEOSCAN)
Brief Title: Neoadjuvant Platinum-based Chemotherapy for Patients With Resectable , Non-small Cell Lung Cancer With Switch to Chemotherapy Alternative in Nonresponders (NEOSCAN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-106
Record Dates: First submitted 2011-09-26; First posted 2011-09-29 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Lung Cancer
Keywords: Carboplatin; Cisplatin; Pemetrexed (Altima); Taxotere (Docetaxel); Vinorelbine Tartrate (Navelbine); Stage IB-III; non squamous; non-small cell lung cancer; 11-106
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Carboplatin; Gemcitabine; Vinorelbine; Docetaxel

ARMS (1):
- pemetrexed plus cisplatin, vinorelbine and docetaxel (Experimental): This is a phase 2 clinical trial for patients with clinical Stage IB-III resectable and operable non-small cell lung cancer, evaluating whether the switch to an alternative, non-platinum neoadjuvant chemotherapy is safe and effective in patients who do not respond to neoadjuvant platinum-based chemotherapy. Those who fail to respond to platinum-based chemotherapy will be switched to the alternative neoadjuvant chemotherapy vinorelbine 45 mg/m2 and docetaxel 45 mg/m2 on day 1 followed by pegylated filgrastim on day 2, repeated every 2 weeks for 4 doses, followed by repeat FDG PET and CT scan.
  Interventions: Drug: pemetrexed; Drug: cisplatin; Drug: Carboplatin; Drug: Gemcitabine Hydrochloride; Drug: Vinorelbine Tartrate; Drug: Docetaxel

INTERVENTIONS:
Drug: pemetrexed
Drug: cisplatin
Drug: Carboplatin
Drug: Gemcitabine Hydrochloride
Drug: Vinorelbine Tartrate
Drug: Docetaxel

SUMMARY:
The purpose of this study is to test a new approach to the use of standard drugs before surgery in patients with lung cancer. This study will find out what effects, good and/or bad, that this approach has on the cancer.

It is routine to give chemotherapy prior to surgery in patients with this type of lung cancer, to help keep it from coming back. It is also routine to perform a special type of scan called a PET scan. This PET scan measures how active a cancer is by use of a special tracer made out of sugar. In this study, all patients will have a PET scan and then be treated with standard chemotherapy drugs, either pemetrexed and cisplatin if the cancer is a "non-squamous" cancer or gemcitabine and cisplatin if the cancer is a squamous cancer. In rare cases, the doctor will decide to give carboplatin instead of cisplatin. In most patients, a repeat PET scan will show that the tumor is decreasing and they will complete standard chemotherapy then go on to have surgery.

In some patients, a repeat PET scan will show that the tumor has not decreased enough. For these patients, the routine practice is to proceed with surgery. This research study will test whether switching from the standard treatment of pemetrexed and cisplatin or gemcitabine and cisplatin to a different treatment called vinorelbine and docetaxel is safe and effective. Vinorelbine and docetaxel are also standard chemotherapy drugs which work in a different way than pemetrexed or gemcitabine and cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of NSCLC at MSKCC
* Stages IB, IIA, IIB, IIIA or IIIB NSCLC
* Primary tumor must measure ≥ 2 cm on CT imaging (per PERCIST guidelines)
* Primary tumor must be FDG-avid with an SUVmax >4.5 (to be consistent with PERCIST guidelines)
* Patients must be candidates for resection with curative intent
* Age ≥ 18 years
* Karnofsky performance status ≥ 70%
* Normal bone marrow function
* leukocytes ≥ 3,000/μl
* absolute neutrophil count ≥ 1,500/μl
* platelets ≥100,000/μl
* hemoglobin ≥9gm/dl.
* Adequate hepatic function
* Total bilirubin ≤1.5 x ULN
* AST ≤ 1.5 x UNL, ALT ≤ 1.5 x ULN
* Alkaline phosphatase ≤ 1.5x ULN
* Women of childbearing age must have a negative pregnancy test
* Men and women of childbearing potential must be willing to use effective contraception while on treatment and for at least 3 months thereafter
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients must not be receiving any other investigational agents
* History of myocardial infarction or unstable angina within the past 12 months Patients with peripheral neuropathy > grade 1
* Other serious illness or medical condition including unstable cardiac disease requiring treatment, history of significant neurologic or psychiatric disorders (including psychotic disorders, dementia, or seizures), or active uncontrolled infection.
* Patients with diabetes mellitus requiring insulin therapy (per PERCIST guidelines)
* Patients with third space fluid which cannot be adequately controlled with drainage
* Women who are pregnant or breast-feeding
* Psychiatric illness or social situation that would limit compliance with study requirements
* Patients with known HIV infection requiring antiretroviral medications and those with AIDS
* Baseline subjective hearing deficit, even if it does not require a hearing aid or intervention, or interfere with activities of daily living (CTCAE grade 2 or higher)
* Baseline renal function <60 ml/min as calculated by the equation of Cockcroft and Gault using the patient's age, weight (kg), and serum creatinine (mg/dl).
* Congestive heart failure with New York Heart Association functional classification > II, characterized by fatigue, dyspnea or other symptoms which limit activities of daily life.

Selection of Pemetrexed versus Gemcitabine: Patients treated with pemetrexed must meet all of the following criteria:

* Non-squamous histology
* Patients must have the ability to interrupt non-steroidal anti-inflammatory drugs (NSAIDs) 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of pemetrexed
* Patients must have the ability to take folic acid, Vitamin B12, and dexamethasone according to protocol
* Patient refuses to take cisplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie E. Chaft, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Patients with clinical Stage IB-III resectable and operable non-small cell lung cancer
Period: Overall Study
Arm/Group | All Patients
Started | 42
Completed | 13
Not Completed | 29
Not completed — Responded to neoadjuvant platinum txt | 27
Not completed — Withdrawal by Subject | 1
Not completed — Patient had brain mets | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: PERCIST Partial Metabolic Response
Description: The primary endpoint was partial metabolic response after 2 cycles of "switch" therapy as assessed by PERCIST (SUVmax decrease ≥30% using the pre-switch scan as new baseline).
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 13
participants | 6

2. Secondary Outcome: Pathologic Response Rate
Description: The percentage of patients with a major pathologic response
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | All Patients
Number analyzed (Participants) | 36
percentage of patients | 17 [6 to 33]

ADVERSE EVENTS:
Description: There was not a comparative toxicity analysis done. CTCAE toxicities were collected for all patients. A comparative toxicity of those patients who switched versus those who did not was not seen as clinically relevant. Hematologic toxicities are anticipated with all chemotherapy.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 4/42
Other Adverse Events (participants affected / at risk) | 34/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=42)
Anorectal infection (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (General disorders) | 1
Febrile neutropenia (General disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Thromboembolic event (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=42)
Hyperglycemia (Metabolism and nutrition disorders) | 23
Hyperglycemia (Metabolism and nutrition disorders) | 13
Neutrophil count decreased (Blood and lymphatic system disorders) | 11
White blood cell decreased (Blood and lymphatic system disorders) | 11
Lymphocyte count decreased (Blood and lymphatic system disorders) | 9
Fatigue (General disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 7
Anemia (Metabolism and nutrition disorders) | 6
Hypertension (Cardiac disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes